CLINICAL TRIAL: NCT04656197
Title: Identification of the Ocular Microbiome and Its Role on Dry Eye Disease
Brief Title: The Ocular Microbiome in Patients With Dry Eye Disease
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2019-01670
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Dry Eye Disease
Keywords: Ocular metagenome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA isolated from eye swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with dry eye disease
  Interventions: Other: Ocular microbiome
- Healthy controls
  Interventions: Other: Ocular microbiome

INTERVENTIONS:
Other: Ocular microbiome — Taxonomical and functional characterization of the ocular microbiome

SUMMARY:
The primary objective of this study is the characterization of the ocular microbiome in a healthy cohort and in patients with dry eye disease using whole-metagenome shotgun sequencing. Secondary objectives are the identification of differences between the ocular microbiome of healthy controls and patients with dry eye disease as well as between the ocular and the gut microbiome.

DETAILED DESCRIPTION:
Dry eye disease is considered to be the most common ocular surface disease worldwide. Recent studies revealed that the ocular microbiome plays an important role in maintaining ocular surface homeostasis and health. Commensals colonizing the ocular surface seem to support the local innate immune system. As the ocular microbiome coordinates several functions together with ocular mucosal and immune epithelial cells, alteration of the microbiome can lead to changes in the integrity of the ocular surface. This can lead to the development of ocular surface related diseases such as dry eye. Inflammation seems to be a key component of dry eye disease in terms of being a propagator as well as a consequence. In contrast to earlier approaches of identifying the microbiome by cultivating with only limited results, it is now possible to provide more details regarding all microbiota residing on the ocular surface due to modern sequencing techniques. Thus, the overall aim of this study is the identification of the role of the ocular microbiome in dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign informed consent
* Patients 60 years of age or older

Exclusion Criteria:

* Patients not willing or able to sign informed consent
* Patients younger than 60 years
* Smoking
* Wearing contact lenses
* Recent (3 month) history of use of systemic and/or topical antibiotics
* Usage of medical eye drops (Lacrycon and other moisturizing eye drops are allowed)
* Recent (3 month) history of ocular surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive ongoing recruitment of subjects attending routine follow-ups through the involved investigators in daily clinical practice at Department of Ophthalmology, Inselspital, Bern
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Characterization of the ocular microbiome | at baseline

SECONDARY OUTCOMES:
Identification of differences of the ocular microbiome between patients and controls | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, Prof. Dr. Dr., Principal Investigator — Department of Ophthalmology, Inselspital, Bern
Locations (1):
- Department of Ophthalmology, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zysset-Burri DC, Schlegel I, Lincke JB, Jaggi D, Keller I, Heller M, Lagache SB, Wolf S, Zinkernagel MS. Understanding the Interactions Between the Ocular Surface Microbiome and the Tear Proteome. Invest Ophthalmol Vis Sci. 2021 Aug 2;62(10):8. doi: 10.1167/iovs.62.10.8. PMID 34369983